CLINICAL TRIAL: NCT01530113
Title: Childhood Sexual Abuse, Vaginismus and Labor Dystocia: Towards a Theoretical Model
Brief Title: Childhood Sexual Abuse, Vaginismus and Labor Dystocia
Acronym: CSA-V-LD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Other Study IDs: -0085-11
Record Dates: First submitted 2012-01-25; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-01

CONDITIONS: Child Abuse; Vaginismus; Dystocia; Depression
Keywords: Childhood sexual abuse; Vaginismus; Partial vaginismus; Labor dystocia; Depression
MeSH Terms: conditions — Vaginismus; Dystocia; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to develop a theoretical model explicating the inter-relationships between Childhood Sexual Abuse (CSA), Partial Vaginismus (PV) and Labor Dystocia (LD), including their associations with Depression (D) as a mediating variable.

The following research hypotheses will be tested:

1. CSA will serve as a risk factor for D, PV and LD.

   * pregnant women with a history of CSA will have higher levels of D compared to pregnant women without a history of CSA.
   * pregnant women with a history of CSA will have more PV compared to pregnant women without a history of CSA.
   * pregnant women with a history of CSA will have higher levels of LD compared to pregnant women without a history of CSA.
2. D will serve as a mediator between prenatal PV and LD.
3. PV will serve as a risk factor for LD.
4. postpartum PV will be affected by childbirth (LD vs. no LD) contingent on the level of D.

DETAILED DESCRIPTION:
Previous studies indicate that childhood sexual abuse has long term implications to women's psychological and physical well-being; among them, depression, a plethora of gynecological symptoms and labor dystocia. Literature in the field also suggests that childhood sexual abuse may be a contributing factor to total and/or partial vaginismus: psycho-sexual disorders associated with significant difficulty and pain during attempted penetration, pelvic examinations and/or sexual relations.

The proposed quantitative longitudinal study aims to develop a theoretical model explicating the relationships between: childhood sexual abuse, prenatal and postpartum partial vaginismus, and childbirth (labor dystocia versus no labor dystocia); including their associations with depression as a mediating variable. Questionnaire responses of pregnant women (Hebrew/Arabic speakers) from the Hillel-Yaffe medical center in Israel will be included in the study.

Data collection will be extended across three time periods: prenatal (third trimester of pregnancy), within one month postpartum, and approximately six months postpartum. Study questionnaires will probe participant's socio-demographic and gynecological history, traumatic life events, sexual experiences, level of depression, partial vaginismus and sexual distress and the objective and subjective severity of their childbirth experience.

Simulations for this project were carried out to help set statistical significance goals and to determine the sample size needed to achieve these goals. From these simulations, a sample size of N=2000 was determined to be adequate and cost effective, to determine standard deviations SD (defining confidence interval ±SD) of about 0.022 for the correlations.

The potential significance of the study is twofold: Theoretically, the study represents a first of its kind effort to explore the relationships between child sexual abuse, prenatal and postpartum partial vaginismus, childbirth and depression, in a single comprehensive longitudinal research study. Practically, the study may potentially assist a wide range of health care professionals by:

1. providing a developing theory for evidence-based practice.
2. showing the need for integration of women's past history into prenatal and postnatal care as a means of lowering the risk for a traumatic birth experience and later psychological distress.
3. aiding in the development of intervention models for the treatment of women with a history of child sexual abuse and/or vaginismus during pregnancy and childbirth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in their third trimester

Exclusion Criteria:

* alcohol addiction
* drug addiction
* mental retardation
* active psychopathology

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women in their third trimester
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Hallak, M.D, Prof., Principal Investigator — Hillel Yaffe Medical Center; Rachel Lev-Wiesel, Ph.D, Prof., Principal Investigator — Haifa University; Hila Sharabi, M.D, Study Director — Hillel Yaffe Medical Center; Ruth Gottfried, Ph.D Student, Study Director — Haifa University
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel